CLINICAL TRIAL: NCT05521321
Title: Feasibility and Acceptability of the Cannabis Awareness and Prevention Toolkit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Bonnie Halpern-Felsher, Marron and Mary Elizabeth Kendrick Professor in Pediatrics II, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 58068; 1R34DA053704 (NIH)
Record Dates: First submitted 2022-08-26; First posted 2022-08-30 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Cannabis Use
Keywords: youth; cannabis; education; health; prevention; marijuana
MeSH Terms: conditions — Marijuana Abuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Receives the Stanford Cannabis Prevention and Awareness curriculum (Experimental): Stanford Cannabis Prevention and Awareness curriculum administered
  Interventions: Behavioral: Stanford Cannabis Awareness and Prevention curriculum
- Does not receive Stanford Cannabis Prevention and Awareness curriculum (No Intervention): Receives another curriculum or no cannabis prevention curriculum

INTERVENTIONS:
Behavioral: Stanford Cannabis Awareness and Prevention curriculum — Stanford Cannabis Awareness and Prevention curriculum delivered as a 5-session course administered in a school classroom setting.
  Arms: Receives the Stanford Cannabis Prevention and Awareness curriculum

SUMMARY:
The Stanford Tobacco Prevention Toolkit is a free, online Toolkit that consists of a curriculum, educational resources, and a resource directory to be used by educators, parents, juvenile justice workers, and healthcare providers to increase knowledge and awareness of cannabis and reduce use among youth. The aim of this study is to investigate the extent to which the curriculum changes students' intentions to use and actual use of cannabis.

ELIGIBILITY:
Inclusion Criteria:

* Middle school and high school students receiving health education at schools participating in the study

Exclusion Criteria:

-

Ages: 10 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 443 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2025-05-16 (Actual); Study Completion 2025-05-16 (Actual)

PRIMARY OUTCOMES:
Change in cannabis use | Change from baseline to follow-up at approximately 156 weeks
  Investigator-originated survey measures (questions) assess ever cannabis use & past 30-day cannabis use. This outcome measure assesses cannabis use.
Change in intention to use cannabis in the future | Change from baseline to follow-up at approximately 156 weeks
  Investigator-originated survey measures (questions) assessing change in participant intention to use cannabis in the future

CONTACTS AND LOCATIONS:
Overall Officials: Bonnie Halpern-Felsher, Ph.D., Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-06-30): https://cdn.clinicaltrials.gov/large-docs/21/NCT05521321/ICF_000.pdf